CLINICAL TRIAL: NCT03478904
Title: Study to Compare Capsule and Liquid Formulations of Enzalutamide After Single Dose Administration Under Fasting Conditions in Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study drug is now commercially available in tablet format
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Figg, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 180070; 18-C-0070
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: Castration Resistant Prostate Cancer; Androgen Receptor
MeSH Terms: conditions — Prostatic Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4x40mg Enzalutamide Capsule Followed by 160mg Enzalutamide Liquid (Experimental): Enzalutamide capsule (Treatment A) followed by enzalutamide liquid (Treatment B)
  Interventions: Drug: Enzalutamide Liquid; Drug: Enzalutamide Capsule
- 160mg Enzalutamide Liquid Followed by 4x40mg Enzalutamide Capsule (Experimental): Enzalutamide liquid (Treatment B) followed by enzalutamide capsule (Treatment A)
  Interventions: Drug: Enzalutamide Liquid; Drug: Enzalutamide Capsule

INTERVENTIONS:
Drug: Enzalutamide Liquid — Enzalutamide liquid formulation given orally (160mg)
  Other Names: ASP-9785
Drug: Enzalutamide Capsule — Enzalutamide gel capsule (4X 40mg)
  Other Names: ASP-9785

SUMMARY:
Background:

Enzalutamide is given to treat metastatic prostate cancer. But it takes 4 pills to deliver the effective dose. This can be difficult for people already taking multiple drugs. And swallowing may be difficult for some people. Researchers want to test out a new way of giving enzalutamide by mouth. They want to see if giving a person the liquid taken from inside the standard 4 gelatin capsules is handled by the body in the same way as giving them the capsules whole.

Objectives:

To compare how capsule and liquid forms of enzalutamide are handled by people with prostate cancer.

Eligibility:

Men at least 18 years old with prostate cancer

Design:

Participants will be screened with a heart test (electrocardiogram), medical history, and physical exam. A tissue sample or lab reports will be reviewed.

During the study, participants will repeat screening tests and have urine tests.

Participants will be randomly assigned to get the study drug in one of two orders: either the as capsules then the liquid form (Arm A) or as the liquid form then the capsule form (Arm B).

Participants will be counseled about birth control.

The study will have 2 periods with a minimum 42 day break in between.

On Day 1 of Period 1 and Day 1 of Period 2, participants will be admitted to the hospital. They will get one dose of the study drug. They cannot eat or drink anything except water for at least 10 hours before and for 4 hours after the study drug. Their blood will be sampled over 24 hours. Lunch and dinner will be served. Participants will answer questions after taking the liquid form.

Participants will have blood drawn on Day 3, Day 8, and Day 42.

DETAILED DESCRIPTION:
Background:

* Enzalutamide is currently approved for the treatment of patients with metastatic castration-resistant prostate cancer (mCRPC)
* The marketed (reference) formulation of enzalutamide is a liquid-filled, soft gelatin capsule containing 40 mg enzalutamide dissolved in Labrasol; four such capsules are required to deliver a 160 mg dose
* The four-capsule regimen is inconvenient because of the number of capsules that must be taken, particularly in light of the fact that cancer patients usually have to take multiple drugs.
* Additionally, some patients may not be able to swallow pills; therefore, alternate methods of oral administration are necessary

Objectives:

-To evaluate the bioequivalence, safety, and tolerability of two oral formulations of enzalutamide following a single 160 mg dose in male subjects with prostate cancer under fasting conditions.

Eligibility:

-Male subjects with prostate cancer

Design:

* Comparative, randomized, open-label, single-dose, 2-way crossover bioavailability, safety and tolerability study
* Subjects will be randomized in Period 1 to one of two sequences: AB or BA. Following a minimum 42-day washout period, subjects will be crossed over in Period 2 to receive the treatment that they did not receive in Period 1.
* Treatment A will be the standard capsule (reference) formulation; Treatment B will be the liquid formulation (test product)
* Blood samples will be collected for pharmacokinetic analysis

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed prostate cancer.

Note: If histopathological documentation is unavailable, a clinical course consistent with prostate cancer is acceptable.

* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Patients must have adequate organ and marrow function as defined below:

  * Hemoglobin greater than or equal to 9 g/dL
  * leukocytes greater than or equal to 3000/mcL
  * absolute neutrophil count greater than or equal to 1500/mcL
  * platelets greater than or equal to 150000/mcL
  * total bilirubin within normal institutional limits
  * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/ alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) less than or equal to X institutional upper limit of normal
  * creatinine within normal institutional limits

OR

--creatinine clearance greater than or equal to 30 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (calculated via Cockcroft-Gault equation)

* Patients must not have other concurrent malignancies (within the past 2 years with the exception of non-melanoma skin cancer and Rai Stage 0 chronic lymphocytic leukemia), in situ carcinoma of any site, or life threatening illnesses, including untreated infection (must be at least 1 week off intravenous antibiotic therapy before beginning enzalutamide).
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Willingness to travel to National Institutes of Health (NIH) for follow-up visits.
* Men age greater than or equal to 18 years of age. Children are excluded because prostate cancer is not common in pediatric populations. Women are not eligible because this disease occurs only in men
* The effects of enzalutamide on the developing human fetus are unknown. For this reason men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) throughout the course of the study and for 3 months after the last dose. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents (in the past 28 days) or herbal medications (within 7 days).
* Patients must not be on enzalutamide within five half-lives before the first planned dose of the study drug or anticipating to start enzalutamide within the next 3 months of the first planned dose of study drug
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to enzalutamide or other agents used in study.
* Clinically significant cardiac disease, e.g. New York Heart Association (NYHA) classes III-IV; uncontrolled angina, uncontrolled arrhythmia or uncontrolled hypertension, myocardial infarction in the previous 6 months as confirmed by an electrocardiogram (ECG).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are taking medications that may alter the metabolism of enzalutamide. This includes the following: strong or moderate cytochrome P450 family 2 subfamily C member 8 (CYP2C8) inhibitors or inducers; strong cytochrome P450 family 3 subfamily A member 4 (CYP3A4) inhibitors or inducers; or Cytochrome P450 2C9 (CYP2C9), 2C19 or 3A4 substrates with a narrow therapeutic index.
* History of seizure, including any febrile seizure, loss of consciousness, or transient ischemic attach, or any condition that may pre-dispose to seizure (e.g. prior stroke, brain arteriovenous malformation, head trauma with loss of consciousness requiring hospitalization).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William D Figg, Pharm.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cordes LM, Schmidt KT, Peer CJ, Chau CH, Redmond E, Francis D, Karzai F, Madan RA, Figg WD. Study to Compare Capsule and Liquid Formulations of Enzalutamide After Single-Dose Administration Under Fasting Conditions in Prostate Cancer. Oncologist. 2021 Sep;26(9):729-e1493. doi: 10.1002/onco.13919. Epub 2021 Aug 14. PMID 34333820
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-C-0070.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled to receive Enzalutamide capsule (Treatment A) followed by enzalutamide liquid (Treatment B)
  Enzalutamide Liquid: Enzalutamide liquid formulation given orally (160mg)
  Enzalutamide Capsule: Enzalutamide gel capsule (4X 40mg)
Period: Overall Study
Arm/Group | 160mg Enzalutamide Liquid Followed by 4x40mg Enzalutamide Capsule
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled to receive Enzalutamide capsule (Treatment A) followed by enzalutamide liquid (Treatment B)
  Enzalutamide Liquid: Enzalutamide liquid formulation given orally (160mg)
  Enzalutamide Capsule: Enzalutamide gel capsule (4X 40mg)
Arm/Group | 160mg Enzalutamide Liquid Followed by 4x40mg Enzalutamide Capsule
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.2 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under Curve (AUC) for the First Period of Administration and Second Period of Administration of Two Formulations of Enzalutamide and the Active Metabolite of Enzalutamide Following a Single 160mg Dose
Description: AUC is the cumulative drug exposure (drug concentration * time) for this single dose over a 42-day sampling period. Participants were randomized to receive Enzalutamide gel capsule 4x40mg (Treatment A) followed by enzalutamide liquid 160mg orally (Treatment B), or Enzalutamide liquid 160mg orally (Treatment B) followed by enzalutamide gel capsule 4x40mg (Treatment A). The difference in the AUCs were calculated following a published non-parametric and noncompartmental approach. A difference of less than 20% difference in the AUC for the test version vs. the standard formulation would permit the two formulations to be considered bioequivalent."
  *The calculated AUC values for N-Desmethyl Enzalutamide of the "4x40mg Enzalutamide Capsule" formulation was influenced by detectable concentrations of N-Desmethyl Enzalutamide (an active metabolite of Enzalutamide) following the 42 Day washout period between the two doses.
Time Frame: Day 42
Population: No participants were enrolled to receive Enzalutamide capsule (Treatment A) followed by enzalutamide liquid (Treatment B).
Measure: Number; unit: AUC ug*h/mL
Groups:
- 160mg Enzalutamide Liquid: Enzalutamide Liquid: Enzalutamide liquid formulation given orally (160mg)
- 4x40mg Enzalutamide Capsule: Enzalutamide Capsule: Enzalutamide gel capsule (4X 40mg)
Arm/Group | 160mg Enzalutamide Liquid | 4x40mg Enzalutamide Capsule
Number analyzed (Participants) | 1 | 1
AUC ug*h/mL
  Day 42 - Enzalutamide | 329.14 | 295.03
  Day 42 - N-Desmethyl Enzalutamide | 617.52 | 529.18

2. Secondary Outcome: Number of Episodes of Grades 1-5 Nausea and Vomiting on 160mg Enzalutamide Liquid Followed by 4x40mg Enzalutamide Gel Capsule
Description: Nausea and vomiting adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe or medically significant but not immediately life-threatening, Grade 4 is life threatening consequences, and Grade 5 is death related to adverse event.
Time Frame: Day 1, 3, 8, and 42
Population: No participants were enrolled to receive Enzalutamide capsule (Treatment A) followed by enzalutamide liquid (Treatment B); Enzalutamide Liquid: Enzalutamide liquid formulation given orally (160mg); Enzalutamide Capsule: Enzalutamide gel capsule (4X 40mg)
Measure: Number; unit: episodes
Groups:
- Grade 1: Grade 1 is mild.
- Grade 2: Grade 2 is moderate.
- Grade 3: Grade 3 is severe or medically significant but not life-threatening.
- Grade 4: Grade 4 is life-threatening consequences.
- Grade 5: Grade 5 is death related to adverse event.
Arm/Group | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
episodes
  Nausea Day 1 | 0 | 0 | 0 | 0 | 0
  Nausea Day 3 | 0 | 0 | 0 | 0 | 0
  Nausea Day 8 | 0 | 0 | 0 | 0 | 0
  Nausea Day 42 | 0 | 0 | 0 | 0 | 0
  Vomiting Day 1 | 0 | 0 | 0 | 0 | 0
  Vomiting Day 3 | 0 | 0 | 0 | 0 | 0
  Vomiting Day 8 | 0 | 0 | 0 | 0 | 0
  Vomiting Day 42 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0
Description: Here is the number of participants with non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence.
Time Frame: Date treatment consent signed to date off study, approximately 7 months and 24 days.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 160mg Enzalutamide Liquid Followed by 4x40mg Enzalutamide Capsule
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Proportion of Participants With Grade 3 Vomiting Compared Between Two Formulations of Enzalutamide at Each Time Point Using Fishers Exact Test
Description: Proportion of participants with Grade 3 vomiting assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0., compared between two formulations of enzalutamide at each time point using Fishers exact test.
Time Frame: Day 1, 3, 8, and 42
Population: This outcome measure was not done. Planned comparisons between the two formulations of enzalutamide at each time point using Fishers exact test were not conducted due to limited study accrual (n=1).
Arm/Group | 160mg Enzalutamide Liquid Followed by 4x40mg Enzalutamide Capsule
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 7 months and 24 days.
Description: No participants were enrolled to receive Enzalutamide capsule (Treatment A) followed by enzalutamide liquid (Treatment B)
  Enzalutamide Liquid: Enzalutamide liquid formulation given orally (160mg)
  Enzalutamide Capsule: Enzalutamide gel capsule (4X 40mg)
Arm/Group | 160mg Enzalutamide Liquid Followed by 4x40mg Enzalutamide Capsule
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 160mg Enzalutamide Liquid Followed by 4x40mg Enzalutamide Capsule (N=1)
Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT03478904/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT03478904/ICF_001.pdf